CLINICAL TRIAL: NCT03855319
Title: SMR/Theta Neurofeedback Training Improves Cognitive Performance and EEG Activity in Elderly With Mild Cognitive Impairment: A Pilot Study
Brief Title: Neurofeedback Improves Cognitive Performance and EEG Activity in Elderly With Mild Cognitive Impairment
Acronym: Neurofeedel
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fabienne Marlats (Other)
Responsible Party: Sponsor-Investigator, Fabienne Marlats, Neuropsychologist, Broca Hospital
Organization: Broca Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: LUS3EEGNF
Record Dates: First submitted 2019-02-25; First posted 2019-02-26 (Actual); Last update posted 2019-02-28 (Actual); Status verified 2019-02

CONDITIONS: Mild Cognitive Impairment
Keywords: Neurofeedback; Electroencephalography; MCI; Alzheimer
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Neurofeedback

STUDY DESIGN:
Intervention Model Description: no randomized, no controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SMR neurofeedback training to MCI (Experimental): A sensorimotor/theta neurofeedback training consisted of 20 individuals sessions, twice a week during 11 weeks maximum. For each subject, NF was planned and conducted by a neuropsychologist experienced in neurophysiology an neurofeedback. Each session lasted 1h10 minutes and was conducted as follows:
  * Preparation and installation of the electrodes, verification of the impedance, adjustement of the calibration.
  * NF training (tasks and video described below)(45minutes)
  * Feedback and debriefing about the session (15 minutes)
  Interventions: Behavioral: SMR neurofeedback training to MCI

INTERVENTIONS:
Behavioral: SMR neurofeedback training to MCI — The intervention consisted to increase the synaptic strengths and sensitivity within this network. Electroencephalography signals for SMR/theta training was recorded at channel Cz according to the international 10-20 system. Theta rhythm was also recorded and, in this case, SMR was stimulated while theta waves were suppressed.A 32 channels system (EEGDigitrcak Biofeedback plus module, Inc Elmiko Medical) was used for the SMR/theta Neurofeedback training.
  Other Names: SMR; neurofeedback

SUMMARY:
This is a non-pharmacological pilot study showing the improvement of a SMR/theta neurofeedback training program on cognitive performance and EEG activity in Elderly with Mild Cognitive Impairment.

DETAILED DESCRIPTION:
Neurofeedback training (NF) as self-regulation method of brain activity, may be beneficial in elderly with mild cognitive impairment. In this pilot study, the investigators studied whether a sensorimotor(SMR)/theta NF training could improve cognitive performance and brain electrical activity in a sample group of elderly patients with mild cognitive impairment. Twenty participants performed an electroencephalography recording, a battery of neuropsychological tests before the neurofeedback training program (T0), following the neurofeedback training program (T1) and 1-month follow-up (T2).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Mild Cognitive Impairment
* education level of 9 years of studies minimum
* righthandedness
* subjective memory complaint confirmed by an informant
* a Mini Mental Status Examination score >20.
* preserve activity of daily living and absence of dementia.

Exclusion Criteria:

* elderly persons who were under guardianship
* resident in nursing facilities
* neurological disease, psychiatric disease
* and involved in another cogniitve intervention.

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-12-15 (Actual); Primary Completion 2018-12-15 (Actual); Study Completion 2018-12-15 (Actual)

PRIMARY OUTCOMES:
Rey Auditory Verbal Learning test | Assessment at baseline, change from baseline to 11 weeks immediately after the NF training and 1 month follow-up
  Assessment of verbal learning in episodic memory, evaluating the ability to encode, combine, store and long-term consolidation process.

SECONDARY OUTCOMES:
Relative power for delta, theta, alpha, sensorimotor and lower beta frequency bands. | Assessment at baseline, change from baseline to 11 weeks immediately after the NF training and 1 month follow-up
  Electroencephalography was recorded and EEG power spectrum was calculated using the fast Fourier transform. The power spectral density was calculated to extract the relative power for each frequency band and estimated as a log-ratio.

CONTACTS AND LOCATIONS:
Overall Officials: anne-Sophie AR Rigaud, Professor, Principal Investigator — Study Principal Investigator

IPD SHARING:
Plan to Share IPD: No